CLINICAL TRIAL: NCT00796796
Title: A Phase I Study of Temsirolimus and Thoracic Radiation in Non-Small Cell Lung Cancer (NSCLC)
Brief Title: Temsirolimus and Radiation for Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 08-1259 / 201012882
Record Dates: First submitted 2008-11-21; First posted 2008-11-24 (Estimated); Last update posted 2013-07-11 (Estimated); Status verified 2013-07

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: Non-small cell lung cancer; temsirolimus; radiation therapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — temsirolimus; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cohort 1 (Starting Dose) (Experimental): Temsirolimus 20 mg IV weekly for 4 weeks
  Radiation therapy will begin on Day 2, one day after the initial dose of temsirolimus. Treatment will consist of daily fractions of 250 cGy, 5 days per week to a total cumulative dose of 3500 cGy for a total of 14 days.
  Interventions: Drug: Temsirolimus; Radiation: Radiation therapy
- Cohort 2 (Experimental): Temsirolimus 25 mg IV weekly for 4 weeks
  Radiation therapy will begin on Day 2, one day after the initial dose of temsirolimus. Treatment will consist of daily fractions of 250 cGy, 5 days per week to a total cumulative dose of 3500 cGy for a total of 14 days.
  Interventions: Drug: Temsirolimus; Radiation: Radiation therapy

INTERVENTIONS:
Drug: Temsirolimus
  Other Names: Torisel
Radiation: Radiation therapy

SUMMARY:
To determine the maximum tolerated dose of the drug temsirolimus given with radiation therapy for patients with non-small cell lung cancer.

DETAILED DESCRIPTION:
Temsirolimus has demonstrated anti-proliferative and anti-angiogenic activity in multiple epithelial cancers, is well-tolerated, has non-overlapping toxicities with radiation, and has been shown to potentiate the effects of radiation in vitro. Locally advanced non-small cell lung cancer is cured in a minority of patients with concurrent chemoradiation but newer agents are needed. In this study temsirolimus will be studied in combination with radiation in a phase I setting to establish safety.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a histologically or cytologically confirmed diagnosis of NSCLC.
* Patients must have an indication for thoracic radiation.
* Because all patients will be receiving radiation therapy to a thoracic mass, they must have radiographically measurable disease to participate.
* Patients may not be candidates for definitive chemoradiation with curative intent.
* Prior treatment of lung cancer (chemotherapy, radiation therapy, and surgery) are allowed if completed at least 4 weeks prior and if all treatment related toxicities are resolved.
* At least 18 years of age.
* Life expectancy of > 12 weeks.
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2.
* Patients must have adequate organ and marrow function as defined below:

  * leukocytes ≥3,000/mcL
  * absolute neutrophil count ≥1,500/mcL
  * platelets ≥100,000/mcL
  * total bilirubin < 1.5
  * AST(SGOT)/ALT(SGPT) ≤2.5 X institutional upper limit of normal
  * creatinine within normal institutional limits OR
  * creatinine clearance ≥60 mL/min/1.73 m2 for patients with creatinine levels above institutional normal
* The effects of temsirolimus on the developing human fetus at the recommended therapeutic dose are unknown. For this reason, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Patients who have had prior treatment with temsirolimus.
* Patients may not be receiving any other investigational agents.
* Patients with symptomatic brain metastases. Known brain metastases are allowed if asymptomatic and previously treated.
* Patients may not be receiving enzyme-inducing antiepileptic drugs (EIAEDs; e.g., phenytoin, carbamazepine, phenobarbital) nor any other CYP3A4 inducer such as rifampin or St. John's wort, as these may decrease temsirolimus levels. A partial list of agents which interact with cytochrome P450 (CYP3A) is found in Appendix B. Use of agents that potently inhibit CYP3A (and hence may raise temsirolimus levels), such as ketoconazole, is discouraged, but not specifically prohibited. Temsirolimus can inhibit CYP2D6, and may decrease metabolism (and increase drug levels) of drugs that are substrates for CYP2D6, such as codeine. The appropriateness of use of such agents is left to physician discretion. A list of drugs that may have potential interactions with CYP2D6 is found in Appendix B. If there is any doubt about eligibility based on concomitant medication, the Principal Investigator should be contacted. All concomitant medications must be recorded.
* Patients with known hypersensitivity reactions to macrolide antibiotics (such as erythromycin, clarithromycin, and azithromycin).
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Known HIV-positive patients on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions. In addition, these patients are at increased risk of lethal infections when treated with marrow-suppressive therapy. Appropriate studies will be undertaken in patients receiving combination antiretroviral therapy when indicated.
* Patients having received prior thoracic radiation therapy directed to the tumor volume to be treated with radiotherapy on this protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2009-03; Primary Completion 2011-06 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Determine the maximum tolerate dose of temsirolimus given with radiation | 90 days after completion of all patients on treatment
  Treatment lasts approximately 4 weeks

SECONDARY OUTCOMES:
Determine the dose limiting toxicities of temsirolimus and radiation in NSCLC patients | 90 days after completion of treatment
  Treatment lasts approximately 4 weeks
Describe phospho-Akt and phospho-S6 levels in circulating mononuclear cells before and after treatment. | Prior to initial temsirolimus dose, one hour post completion of initial temsirolimus dose, and prior to second temsirolimus dose
Safety of the regimen in patients with NSCLC | 90 days after completion of treatment
  Treatment lasts approximately 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Maria Q. Baggstrom, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

REFERENCES:
- [Background] Hudes G, Carducci M, Tomczak P, Dutcher J, Figlin R, Kapoor A, Staroslawska E, Sosman J, McDermott D, Bodrogi I, Kovacevic Z, Lesovoy V, Schmidt-Wolf IG, Barbarash O, Gokmen E, O'Toole T, Lustgarten S, Moore L, Motzer RJ; Global ARCC Trial. Temsirolimus, interferon alfa, or both for advanced renal-cell carcinoma. N Engl J Med. 2007 May 31;356(22):2271-81. doi: 10.1056/NEJMoa066838. PMID 17538086
- [Background] Schmelzle T, Hall MN. TOR, a central controller of cell growth. Cell. 2000 Oct 13;103(2):253-62. doi: 10.1016/s0092-8674(00)00117-3. PMID 11057898
- [Background] Williams KJ, Telfer BA, Xenaki D, Sheridan MR, Desbaillets I, Peters HJ, Honess D, Harris AL, Dachs GU, van der Kogel A, Stratford IJ. Enhanced response to radiotherapy in tumours deficient in the function of hypoxia-inducible factor-1. Radiother Oncol. 2005 Apr;75(1):89-98. doi: 10.1016/j.radonc.2005.01.009. Epub 2005 Apr 18. PMID 15878106
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu